CLINICAL TRIAL: NCT00509782
Title: Phase I Trial of ZIO-101 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0909
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; Anti-Tumor Effects; ZIO-101
MeSH Terms: interventions — darinaparsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZIO-101 (Experimental)
  Interventions: Drug: ZIO-101

INTERVENTIONS:
Drug: ZIO-101 — Starting Dose 78 mg/m^2 intravenously daily for 5 consecutive days repeated every 4 weeks.

SUMMARY:
Primary Objectives:

1. To determine the toxicities and maximum tolerated dose (MTD) of ZIO-101 when administered intravenously once a day for 5 consecutive days every 4 weeks in subjects with advanced solid tumors.
2. To determine the pharmacokinetic profile of ZIO-101 when administered intravenously once a day for 5 consecutive days every 4 weeks.

Secondary Objective:

1. To determine the anti-tumor effects of ZIO-101.

DETAILED DESCRIPTION:
ZIO-101 is a drug that may change cancerous cells into healthy (benign) cells. It is also designed to cause cancer cells to destroy themselves; a term called apoptosis.

Before you can start treatment on this study, you will have what are called "screening tests" no more than one week before starting the study. These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete medical history and physical exam, including measurements of your weight, blood pressure, pulse, and temperature. You will also be asked what other medicines you are taking and about your general well-being. You will have an electrocardiogram (ECG - a test to measure the electrical activity of the heart). Blood (about 2 1/2 tablespoons) will be drawn. A sample of urine will be also be collected and tested to see if your kidneys are working correctly. Women who are able to have children must have a negative urine pregnancy test.

To see the current condition of your tumor, additional tests may need to be performed if they have not already been done recently. These tests may include a chest x-ray, a CT scan (imaging computer pictures of your body), a bone scan (an imaging test of your bones with a contrast material), or an MRI (a detailed imaging scan of certain areas of your body).

If you are found to be eligible to take part in this study, you will begin treatment with ZIO-101. Immediately before being treated with ZIO-101 on Day 0, you will have another physical exam and you will be asked about any medicines you are taking and how you are feeling. You will also be asked a series of questions which will assess your mental health. This is called a mini-mental status exam and will take approximately 10 minutes to complete. The blood tests may need to be repeated along with the ECG and the urine test. In addition, a small blood sample (about 10 teaspoons) must be taken immediately before the injection of ZIO-101. This blood will be used to help in the measurement of drug levels in the blood. These are called pharmacokinetic (PK) tests. This blood sample will also be used to measure arsenic levels in your blood.

ZIO-101 will be injected into your vein over 60 minutes in the clinical translational research center of UTMDACC. This drug must be given through a special IV called a central line catheter so that it does not damage your surrounding tissue. You will have to sign a separate consent document before placement of a catheter can be performed. Special care will be taken to be sure the drug does not leak into surrounding tissue. The use of anti-nausea and other supportive care medications may be given during the infusion.

Following the injection, you will have 6 samples of blood taken for PK tests at half an hour and 1, 2, 4, 8, and 12 hours after finishing the treatment.

For the next 4 days at about the same time as your first infusion, you will be prepared for treatment with ZIO-101. Before each injection, you will be asked how you feel, an ECG will be performed, and a small sample of blood (about 2 teaspoons) will be drawn for PK tests. The Day 1-4 infusions will also each take about 1 hour. In total you will receive 5 daily injections of ZIO-101. On Day 4 at the end of the infusion, another sample of blood will be drawn (about 5 teaspoons) to measure arsenic levels in your blood.

Your next visit will be Week 2 and at the start of this visit, a blood sample (about 2 teaspoons) will be drawn for PK tests, and you will be asked how you feel. At Week 3, another blood sample (about 7 teaspoons) will be drawn for PK tests, and to measure arsenic levels in your blood, and you will again be asked how you feel.

At Week 4, a new cycle begins. Immediately before being treated with ZIO-101, you will have a physical examination and you will take a mini-mental status examination; you will be asked about any medicines you are taking and how you are feeling. The blood tests will be repeated along with the ECG and the routine urine test. In addition, tests to measure your tumor will be repeated.

This study is trying to find the best dose of ZIO-101. At first, 3 patients will be assigned to the first dose level. They will be followed to evaluate their side effects for a period of 4 weeks before 3 more patients are enrolled. If none of the patients develop serious side effects, the dose escalation will continue. If 1 of the 3 patients in a particular dose level develops significant side effects, 3 more patients will be enrolled at that level. If 2 or more of the 6 patients develop serious side effects, then the escalation will finish and all future patients on this study will be treated at a lower dose level (half way between this level and the previous one).

You may receive up to 6 cycles of treatment. You may be taken off study early if your disease gets worse or intolerable side effects occur. Once you go off study, you will have an end of study visit. During this visit, you will have a physical exam, a mini-mental status exam and blood (about 3 teaspoons) will be drawn for routine tests.

This is an investigational study. ZIO-101 has been authorized by the FDA for use in research only. ZIO-101 will be provided free of charge during the study. Also, any tests or procedures that are being done solely for the purpose of this research study will be provided free of charge. Up to 50 patients will take part in this multicenter study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmation solid malignancy refractory to conventional standard therapies for their condition.
2. Eligible subjects MUST have at least one measurable lesion as defined by RECIST guidelines. If the measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology. Measurable lesions MUST not have been in a previously irradiated field or injected with biological agents.
3. Pediatric patients will be eligible at the discretion of the primary investigator.
4. ECOG performance status score </= 2.
5. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use acceptable contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative blood or urine pregnancy test within 1 week before beginning treatment. Sexually active men must also use acceptable contraceptive methods.
6. Patients must provide written informed consent prior to treatment.
7. At least four weeks from completion of prior therapy to day 1 of study drug.
8. Baseline toxicity assessment less than or equal to grade 1 except treatment induced alopecia (NCI Common Terminology Criteria for Adverse Events [CTCAE] version 3.0).
9. Evidence of adequate multi-organ functional status as reflected by the following clinical laboratory values: - Serum creatinine </= 2 times the upper normal limit OR a calculated creatinine clearance </= 50 cc/min. - Total bilirubin </= 2 times the upper normal limit. - Alanine aminotransferase (ALT), OR aspartate aminotransferase (AST) </= 3 times the upper limit of normal.
10. Granulocytes in peripheral blood greater than or equal to 1 x 10(9) per liter, hemoglobin greater than or equal to 8.5 g/dL, and platelets greater than or equal to 50,000 cells/microL.

Exclusion Criteria:

1. Uncontrolled systemic infection (documented with microbiological studies).
2. Active heart disease as defined by an acute myocardial infarction within the previous 6 months before starting therapy, stable or unstable angina, clinically significant arrhythmia requiring medical management, OR New York Heart Association Classification of Functional Activities. Class 3: Patient has marked limitation in activities due to symptoms, even during less-than-ordinary activity and is comfortable only at rest OR Class 4: Severe limitations. Patient experiences symptoms even while at rest.
3. Concomitant therapy for solid cancer.
4. Pregnant subjects and those who are breast-feeding.
5. History of an invasive second primary malignancy diagnosed within the previous 3 years except for Stage I Endometrial/Cervical Carcinoma or Prostate Carcinoma treated surgically, and non-melanoma skin cancer.
6. Documented personal or family history of prolonged QT syndrome.
7. 12 lead electrocardiogram with a corrected QT interval >/= 460 milliseconds.
8. History of confusion or dementia.
9. History of seizure disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Daily for 5 consecutive days repeated every 4 weeks for 1 cycle; evaluation of 4-6 dose escalations to determine an MTD

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Tsimberidou AM, Camacho LH, Verstovsek S, Ng C, Hong DS, Uehara CK, Gutierrez C, Daring S, Stevens J, Komarnitsky PB, Schwartz B, Kurzrock R. A phase I clinical trial of darinaparsin in patients with refractory solid tumors. Clin Cancer Res. 2009 Jul 15;15(14):4769-76. doi: 10.1158/1078-0432.CCR-08-2984. Epub 2009 Jul 7. PMID 19584162
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org